CLINICAL TRIAL: NCT00454701
Title: Assessment and Tracking of Long-term Alefacept (LFA-3/IgG1 Fusion Protein) Safety (ATLAS)
Brief Title: Assessment and Tracking of Long-term Alefacept Safety
Acronym: ATLAS
Status: Terminated | Type: Observational
Why Stopped: The Sponsor has made a decision, driven by business needs, to cease promotion, manufacturing, distribution and sales of Amevive
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: 0485-CL-0001; C-736
Record Dates: First submitted 2007-03-29; First posted 2007-04-02 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-12

CONDITIONS: Psoriasis
Keywords: Psoriasis; Alefacept; Amevive®; Drug exposure
MeSH Terms: conditions — Psoriasis | interventions — Alefacept

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1. Amevive Exposure: Patients treated with alefacept for chronic plaque psoriasis
  Interventions: Drug: Alefacept exposure

INTERVENTIONS:
Drug: Alefacept exposure — Observational
  Other Names: Amevive; ASP0485

SUMMARY:
Subjects exposed to alefacept are to be enrolled. Subjects will be contacted every 6 months to gather general health information.

DETAILED DESCRIPTION:
There are no study-mandated tests, visits or clinical interventions after the 1st (enrolling) visit. After the patient is enrolled in the study, they will be contacted every 6 months to complete structured telephone interviews conducted by the ATLAS Study Center.

ELIGIBILITY:
Inclusion Criteria:

* Psoriasis patients who are prescribed alefacept consistent with product labeling are eligible for enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with alefacept for chronic plaque psoriasis
Sampling Method: Non-Probability Sample
Enrollment: 1897 (Actual)
Dates: Start 2003-06; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
To measure the rates of non-Hodgkin's lymphoma (NHL) and infections that require hospitalization occurring in psoriasis patients treated with alefacept | At six month intervals for five years

SECONDARY OUTCOMES:
To estimate the rates of lung cancer, breast cancer (female), prostate cancer, colorectal cancer, melanoma and active tuberculosis within a population of patients with psoriasis treated with alefacept. | At six month intervals for five years

CONTACTS AND LOCATIONS:
Overall Officials: Vice President Medical Affairs, Study Director — Astellas Pharma Global Development
Locations (268):
- United States (241):
  - Total Skin and Beauty Dermatology Center, Birmingham, Alabama
  - Janet Cash, Birmingham, Alabama
  - Bay Shore Dermatology & Laser Surgery Center, Fairhope, Alabama
  - Eric Baum, Gadsden, Alabama
  - Ruth A Yates, Huntsville, Alabama
  - Mobile Dermatology, Mobile, Alabama
  - English Dermatology Centers, Phoenix, Arizona
  - Scottsdale Dermatology, Scottsdale, Arizona
  - Sheftel & Associates Dermatology, Tucson, Arizona
  - Ozark Dermatology Clinic, Fayetteville, Arkansas
  - Cyril E Severns, Fort Smith, Arkansas
  - Burke Pharmaceutical Research, Hot Springs, Arkansas
  - Little Rock Dermatology Clinic, Little Rock, Arkansas
  - East Bay Dermatology Medical Group Inc. DBA Center for Dermatology, Cosmetic & Laser Surgery, Inc, Fremont, California
  - East Bay Dermatology Medical Group Inc., DBA Center for Dermatology, Cosmetic and Laser Surgery, Fremont, California
  - Minarets Medical Group, Inc., Fresno, California
  - John J. Guagenti, MD, Glendale, California
  - Scripps Clinic, La Mesa, California
  - Fairmont Dermatology, Lodi, California
  - California Skin Institute, Mountain View, California
  - Clinical Research Specialists, Inc., Santa Monica, California
  - Advanced Dermatology, Centennial, Colorado
  - Dermatology & Laser Center at Harvard Park, PLLC, Denver, Colorado
  - D.B.A. Colorado West Dermatology, Grand Junction, Colorado
  - Jeremy Moss, MD, Bridgeport, Connecticut
  - Eric R. Wolf, MD, Groton, Connecticut
  - Bender and Kolenik MD, PC, Norwalk, Connecticut
  - Charles Halasz, Norwalk, Connecticut
  - Stuart Bender, Norwalk, Connecticut
  - Jeffrey Alter, Waterbury, Connecticut
  - Panzer Dermatology Assoc., Newark, Delaware
  - Atlantic Skin and Cosmetic Surgery- P.C., Wilmington, Delaware
  - Jerri L. Johnson MD, PA, Altamonte Springs, Florida
  - Center for Dermatology, Boca Raton, Florida
  - Jodi Fiedler, Boca Raton, Florida
  - Dermatology and Skin Surgery Center, PA, Celebration, Florida
  - Brent M Schillinger, Delray Beach, Florida
  - A.G.A. Clinical Trials, Hialeah, Florida
  - North Florida Dermatology Associates, P.A., Jacksonville, Florida
  - Coastal Dermatology, PA, Jacksonville, Florida
  - A Center for Dermatology, Cosmetic and Laser Surgery, Jupiter, Florida
  - Associates in Medical and Surgical Dermatology, Naples, Florida
  - Dermatology & Laser Center, Orange Park, Florida
  - Reflections Dermatology & Center for Skin Care, Orlando, Florida
  - John L. Meisenheimer, MD, Orlando, Florida
  - Advanced Dermatology, Orlando, Florida
  - Ormond Beach Dermatology, Ormond Beach, Florida
  - Waters Edge Dermatology, Palm Beach Gardens, Florida
  - Mark Cheiken, Palm Coast, Florida
  - Timothy Kelly, MD, PA, Palm Harbor, Florida
  - Snyder & Le M.D. PA, Pembroke Pines, Florida
  - Kevin L Welch, Pensacola, Florida
  - Hecker Dermatology Group PA, Pompano Beach, Florida
  - Michael A. Scannon MD, PA, Tampa, Florida
  - Luis T. Menendez, MD, PA, Tampa, Florida
  - Neil S. Heskel, MD, Vero Beach, Florida
  - Sunnycoast Dermatology, Vero Beach, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - Darren Casey, Atlanta, Georgia
  - Georgia Skin Specialists, Atlanta, Georgia
  - Peachtree Dermatology Associates, Atlanta, Georgia
  - Family Dermatology-Cynthia A. Abbott, MD, Atlanta, Georgia
  - Allen B. Filstein, MD, Conyers, Georgia
  - East Metro Dermatology, PC, Conyers, Georgia
  - North Atlanta Dermatology, Duluth, Georgia
  - Dermatologic Surgery Specialist Inc., Macon, Georgia
  - Paul S. Takiguchi- MD- Inc., ‘Aiea, Hawaii
  - Saltzer Medical Group, PA, Nampa, Idaho
  - Altman Dermatology Associates, Arlington Heights, Illinois
  - Thomas Brander, Bloomington, Illinois
  - Calumet Dermatology Associates S.C., Calumet City, Illinois
  - Christie Clinic, Champaign, Illinois
  - Danilo Del Campo, Chicago, Illinois
  - Michael A. Greenberg, MD, Ltd., Elk Grove Village, Illinois
  - North Suburban Dermatology Associates, Gurnee, Illinois
  - Dermatology Associates of LaGrange, LaGrange Highlands, Illinois
  - Soderstrom Dermatology Center, Peoria, Illinois
  - David Coynik, Peru, Illinois
  - Schaumburg Dermatology, Schaumburg, Illinois
  - Alan E. Lasser MD PC, Skokie, Illinois
  - Paul Getz, West Dundee, Illinois
  - Advanced Dermatology Associates, PC, Bloomington, Indiana
  - Spencer Dermatology Associates LLC, Crawfordsville, Indiana
  - Mitchell Bressack, Crown Point, Indiana
  - Fort Wayne Dermatology, Fort Wayne, Indiana
  - Tsu-Yi Chuang, Indianapolis, Indiana
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - Randall Dermatology, West Lafayette, Indiana
  - Timothy Abrahamson, Urbandale, Iowa
  - Dermatology Associates, Waterloo, Iowa
  - Great Plains Dermatology- P.A., Hays, Kansas
  - American Dermatology Associates, Shawnee, Kansas
  - Kansas Medical Clinic, PA, Topeka, Kansas
  - Moeller Dermatology, LLC, Wichita, Kansas
  - Melissa Knuckles, Corbin, Kentucky
  - LA Dermatology Assoc LLC, Baton Rouge, Louisiana
  - Dimitri Dermatology, Gretna, Louisiana
  - Eileen Ringel, Waterville, Maine
  - Benjamin Bernstein, Bel Air, Maryland
  - The Dermatology Group LLC, Chevy Chase, Maryland
  - Dermatology & Advanced Skin Care, Ellicott City, Maryland
  - Greater Washington Dermatology P.A., Rockville, Maryland
  - Todd Colonna, Rockville, Maryland
  - Northeast Dermatology, Beverly, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Bruce Goldstein, Florence, Massachusetts
  - Mark Lewis, Marblehead, Massachusetts
  - Jay A. Goldstein, MD, Natick, Massachusetts
  - Kenneth M. Reed, MD, Quincy, Massachusetts
  - Ronald S. Nadel, Springfield, Massachusetts
  - Wendy McFalda, DO, Clarkston, Michigan
  - Drs. Iacobelli & DiGregorio, PC, Clinton Township, Michigan
  - Psoriasis and Eczema Treatment Center of Western Michigan, Grand Rapids, Michigan
  - Livonia Dermatology, PLLC, Livonia, Michigan
  - Somerset Skin Centre, Troy, Michigan
  - Midwest Center for Dermatology and Cosmetic Surgery, Warren, Michigan
  - Michael T. Siegel MD- P.C., Waterford, Michigan
  - Jeffrey N Samuelson, Burnsville, Minnesota
  - Advancements In Derm, Edina, Minnesota
  - Jack C. Scott, Fridley, Minnesota
  - Steven E. Prawer, Fridley, Minnesota
  - The Dermatology Clinic- PLLC, Gulfport, Mississippi
  - Mark Gallardo, Hattiesburg, Mississippi
  - Andrew Berg, Kansas City, Missouri
  - Sharon K Tiefenbrunn, St Louis, Missouri
  - Associated Dermatology, Helena, Montana
  - Johnnie M Woodson, Las Vegas, Nevada
  - Las Vegas, Nevada
  - Robert B. Stromling, MD, Las Vegas, Nevada
  - Nashua Dermatology Associates, Nashua, New Hampshire
  - Psoriasis Treatment Center of Central NJ, East Windsor, New Jersey
  - North Bergen Dermatologic Group, Ridgewood, New Jersey
  - Buffalo Medical Group, Buffalo, New York
  - Bruce S. Stein, Flushing, New York
  - Advanced Dermatology, Fresh Meadows, New York
  - Frank De Mento, Garden City, New York
  - Garden City Dermatology, P.C., Garden City, New York
  - Edmund Lee, Huntington, New York
  - Jeffrey P Schachne, Jefferson Valley, New York
  - Atlantic Dermatologic Associates, LLC, Lynbrook, New York
  - Orange Dermatology Assoc, PC, Monroe, New York
  - Peter S. Halperin's Office, New York, New York
  - Peter Accetta, Orchard Park, New York
  - Dermatology Partners of Western New York, Rochester, New York
  - Dermatique Dermedy Dermatology- PC, Smithtown, New York
  - Marina I Peredo, MD, Smithtown, New York
  - Josiane Lederman, MD, PC, Staten Island, New York
  - Joseph D. Sutton, MD, Suffern, New York
  - Susan E. Katz MD, The Bronx, New York
  - Martin Morell, MD, Utica, New York
  - Stanley A. Newfield, Valley Stream, New York
  - Alan B Schliftman, White Plains, New York
  - Colleen Demers, Williamsville, New York
  - Lynn A. Amarante, MD PC, Williamsville, New York
  - Davie Dermatology, Advance, North Carolina
  - Skyland Dermatology and Psychiatry, Asheville, North Carolina
  - Curtis W. Schupbach- MD, Charlotte, North Carolina
  - Andrus & Associates Dermatology, PA, Raleigh, North Carolina
  - Atlantic Dermatology Associates, P.A., Wilmington, North Carolina
  - WHA Medical Clinic PLLC, Wilmington, North Carolina
  - William S. Mirando, MD, LLC, Ashtabula, Ohio
  - Eugene Conte, Centerville, Ohio
  - University Dermatology Consultants, Inc., Cincinnati, Ohio
  - Martha Hickmann, MD, Dayton, Ohio
  - Joyce Lender, Elyria, Ohio
  - Northeast Dermatology & Cosmetic Surgery, Gahanna, Ohio
  - Judith Andreano, Strongsville, Ohio
  - Harvey L. Handler, MD, Sylvania, Ohio
  - Medical College of Ohio, Toledo, Ohio
  - Options Health Research, Tulsa, Oklahoma
  - Allergy, Asthma & Dermatology Research Centers, LLC, Lake Oswego, Oregon
  - Eric Olson, Springfield, Oregon
  - Paul Klas, Tualatin, Oregon
  - Robert M. Stiegel- M.D. LTD, Beaver, Pennsylvania
  - Lehigh Valley Dermatology, Bethlehem, Pennsylvania
  - Jan Brydon, Erie, Pennsylvania
  - David Amato, Harrisburg, Pennsylvania
  - Saye & Gette Dermatology Associates, PC, Harrisburg, Pennsylvania
  - Chad Mathews, Hermitage, Pennsylvania
  - Dermatology Associates of Lancaster, Lancaster, Pennsylvania
  - Stephanie Mackey, Lancaster, Pennsylvania
  - Allegheny Dermatology Assoc., PC, Monroeville, Pennsylvania
  - East Penn Dermatology, North Wales, Pennsylvania
  - Paddington Testing Co, Inc., Philadelphia, Pennsylvania
  - Louis H. Martone, MD, PC, Pittsburgh, Pennsylvania
  - Neil M. Niren MD, Pittsburgh, Pennsylvania
  - Dermatology Associates of Plymouth Meeting- P.C., Plymouth Meeting, Pennsylvania
  - Joseph Bikowski, Sewickley, Pennsylvania
  - Joel Seigel- MD, Washington, Pennsylvania
  - Sabrina Dowd, Williamsport, Pennsylvania
  - Clinical Partners, LLC, Johnston, Rhode Island
  - Paul T. Zaydon MD, Pawtucket, Rhode Island
  - Dermatology Associates of the Low Counties, Beaufort, South Carolina
  - Marta Hampton, Charleston, South Carolina
  - Rheumatology Associates, Charleston, South Carolina
  - The Dermatology Group, LLC, Columbia, South Carolina
  - McClerklin Skin and Laser Center, Columbia, South Carolina
  - John Humeniuk, Greenville, South Carolina
  - Lesly S. Davidson MD PA, Mt. Pleasant, South Carolina
  - Grand Strand Dermatology, LLC, Myrtle Beach, South Carolina
  - Hillcrest Dermatology Center, PA, Orangeburg, South Carolina
  - DeVore Dermatology, PA, Spartanburg, South Carolina
  - Palmetto Dermatology, PA, West Columbia, South Carolina
  - Midsouth Dermatology and Skin Cancer Center, Bartlett, Tennessee
  - Advanced Skin & Laser Center, Brentwood, Tennessee
  - Rivergate Dermatology Research Center, Goodlettsville, Tennessee
  - Dermatology Associates of Kingsport, PC, Kingsport, Tennessee
  - Dermatology Associates of Knoxville, PC, Knoxville, Tennessee
  - Delta Medical Ctr., Memphis, Tennessee
  - Abigail James, NP, MSN, Nashville, Tennessee
  - Tennessee Clinical Research Center, Nashville, Tennessee
  - Derm & Skin Cancer Surgery Center, Allen, Texas
  - Arlington Center for Dermatology, Arlington, Texas
  - Bellaire Dermatology Associates, Bellaire, Texas
  - Alpha Therapy Center, Corpus Christi, Texas
  - Raymond Blackburn, Dallas, Texas
  - Betty J. Rajan, Fort Worth, Texas
  - Lisa Garner, Garland, Texas
  - West Houston Dermatology, PA, Houston, Texas
  - Lone Star Children's Medical PLLC, Houston, Texas
  - Dermatology and Laser Center, Irving, Texas
  - Steven J. Smith, MD, Kingwood, Texas
  - Mark S Wallis, Longview, Texas
  - Lubbock Dermatology and Skin Cancer Center, Lubbock, Texas
  - Dermatology of East Texas, Lufkin, Texas
  - Ashkan Ghorbani, Pasadena, Texas
  - Gregory W Thompson, San Antonio, Texas
  - Dermatology Research Associates of Tyler, Tyler, Texas
  - Rocky Mountain Dermatology, Logan, Utah
  - Aspen Clinical Research, LLC, Orem, Utah
  - Four Seasons Dermatology, South Burlington, Vermont
  - Georgia A Seely, Richmond, Virginia
  - Virginia Beach Dermatology Associates, PPLC, Virginia Beach, Virginia
  - Dermatology & Laser Center Northwest, Bellingham, Washington
  - Dermatology Associates, PLLC, Seattle, Washington
  - James Hu MD PC, Seattle, Washington
  - James M. Komorous MD PS, Tacoma, Washington
  - Eastern Washington Dermatology, Walla Walla, Washington
  - Layton Avenue Dermatology, Greenfield, Wisconsin
  - Aylesworth Dermatology SC, Rhinelander, Wisconsin
  - Cheyenne Dermatology- P.C., Cheyenne, Wyoming
- Canada (27):
  - Winnipeg Clinic, Winnepeg, Manitoba
  - Dermadvances Research, Winnipeg, Manitoba
  - Douglas N. Keeling MD Dermatologist PC, Quispamsis, New Brunswick
  - Nexus Clinical Research, St. John's, Newfoundland and Labrador
  - St. John's, Newfoundland and Labrador
  - NewLab Clinical Research, Inc., St. John's, Newfoundland and Labrador
  - Sudbury Skin Clinic, Greater Sudbury, Ontario
  - Dermatrials Research, Hamilton, Ontario
  - Limestone Dermatology & Laser Clinic, Kingston, Ontario
  - Mediprobe Research, Inc., London, Ontario
  - The Guenther Dermatology Research Centre, London, Ontario
  - Wellington Dermatology Associates, London, Ontario
  - Lynderm Research, Inc., Markham, Ontario
  - John J. Turner, MD, Newmarket, Ontario
  - A.M. Katz Medicine D.C., Newmarket, Ontario
  - Dermatology Clinic, North York, Ontario
  - Skin Centre for Dermatology, Peterborough, Ontario
  - Dermatology Associates, Toronto, Ontario
  - Specialized Dermatology, Welland, Ontario
  - Clinique de dermatologie Dr. Francois Bouchard, Alma, Quebec
  - Francoise Giard, Gatineau, Quebec
  - Innovaderm Research, Inc, Montreal, Quebec
  - Siena Medical Research, Montreal, Quebec
  - Giles P. Raymond, Pierrefonds, Quebec
  - CRCMR Gilbert Inc., Québec, Quebec
  - (CRDQ) Centre De Recherche Dermatologique Du Quebec Metropolitan, Québec, Quebec
  - Victoria East Medical Clinic, Regina, Saskatchewan